CLINICAL TRIAL: NCT02143466
Title: A Multi-arm, Phase Ib, Open-Label, Multicentre Study to Assess the Safety,Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of AZD9291 in Combination With Ascending Doses of Novel Therapeutics in Patients With EGFRm+ Advanced NSCLC Who Have Progressed Following Therapy With an EGFR TKI (TATTON).
Brief Title: AZD9291 in Combination With Ascending Doses of Novel Therapeutics
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5160C00006; 2016-004752-29 (EudraCT Number)
Record Dates: First submitted 2014-05-09; First posted 2014-05-21 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Advanced Non Small Cell Lung Cancer
Keywords: Phase I; Safety; Tolerability; Efficacy; Anti-tumour; AZD9291; AZD6094; MEDI4736; Osimertinib; Savolitinib; Selumetinib; Durvalumab; Ascending Doses; Expansion cohorts; EGFR; Advanced Non-Small Cell Lung Cancer; Tyrosine Kinase Inhibitors
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; osimertinib; AZD 6244; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- AZD6094 (Experimental): AZD9291 in combination with AZD6094
  Interventions: Drug: Part A - AZD9291 in combination with AZD6094; Drug: Part B - AZD9291 in combination with AZD6094; Drug: Part C - AZD9291 in combination with AZD6094 (Japan only); Drug: Part D - AZD9291 in combination with AZD6094
- Selumetinib (Experimental): AZD9291 in combination with selumetinib
  Interventions: Drug: Part A - AZD9291 in combination with continuous selumetinib (Asian subjects); Drug: Part A - AZD9291 in combination with continuous selumetinib (non-Asian subjects); Drug: Part A - AZD9291 in combination with intermittent selumetinib; Drug: Part B - AZD9291 in combination with selumetinib
- MEDI4736 (Experimental): AZD9291 in combination with MEDI4736. Enrolment into the patient cohort that evaluated AZD9291 treatment in combination with MEDI4736 as 1st line treatment has been terminated due to an increased incidence of ILD-like events (interstitial lung disease/pneumonitis), and is no longer being evaluated in this study.
  Interventions: Drug: Part A - AZD9291 in combination with MEDI4736; Drug: Part B - AZD9291 in combination with MEDI4736
- AZD6094 (monotherapy) (Experimental): AZD6094 in monotherapy (for Japan only)
  Interventions: Drug: Part C - AZD6094 monotherapy (Japan only)

INTERVENTIONS:
Drug: Part A - AZD9291 in combination with AZD6094 — Part A - AZD9291 and AZD6094 administered in different doses to investigate the safety and tolerability of this combination and define the combination dose for further clinical evaluation in Part B.
  Other Names: Osimertinib & Savolitinib/Volitinib
  Arms: AZD6094
Drug: Part A - AZD9291 in combination with continuous selumetinib (Asian subjects) — Part A - AZD9291 and selumetinib (continuous treatment) administered in different doses to investigate the safety and tolerability of this combination in Asian subjects and to define the combination dose for further clinical evaluation in Part B.
  Other Names: Osimertinib & ARRY-142886
  Arms: Selumetinib
Drug: Part A - AZD9291 in combination with continuous selumetinib (non-Asian subjects) — Part A - AZD9291 and selumetinib (continuous treatment) administered in different doses to investigate the safety and tolerability of this combination in non-Asian subjects and to define the combination dose for further clinical evaluation in Part B.
  Other Names: Osimertinib & ARRY-142886
  Arms: Selumetinib
Drug: Part A - AZD9291 in combination with intermittent selumetinib — Part A - AZD9291 and selumetinib (intermittent treatment) administered in different doses to investigate the safety and tolerability of this combination and to define the combination dose for further clinical evaluation in Part B.
  Other Names: Osimertinib & ARRY-142886
  Arms: Selumetinib
Drug: Part A - AZD9291 in combination with MEDI4736 — Part A - AZD9291 and MEDI4736 administered in different doses to investigate the safety and tolerability of this combination and to define the combination dose for further clinical evaluation in Part B.
  Note: Enrolment into the patient cohort that evaluated AZD9291 treatment in combination with MEDI4736 as 1st line treatment has been terminated due to an increased incidence of ILD-like events (interstitial lung disease/pneumonitis), and is no longer being evaluated in this study.
  Other Names: Osimertinib & Durvalumab
  Arms: MEDI4736
Drug: Part B - AZD9291 in combination with AZD6094 — Part B - AZD9291 and AZD6094 administered in the dose identified in Part A (AZD9291 80mg OD + AZD6094 600mg OD) to further investigate the safety and tolerability of this combination.
  Other Names: Osimertinib & Savolitinib/Volitinib
  Arms: AZD6094
Drug: Part B - AZD9291 in combination with selumetinib — Part B - AZD9291 and selumetinib administered in the dose identified in Part A (AZD9291 80mg OD + selumetinib 75 mg BD intermittent [4 days on/3 days off]) to further investigate the safety and tolerability of this combination.
  Other Names: Osimertinib & ARRY-142886
  Arms: Selumetinib
Drug: Part B - AZD9291 in combination with MEDI4736 — Part B - AZD9291 and MEDI4736 administered in the dose identified in Part A to further investigate the safety and tolerability of this combination.
  Note: Enrolment into the patient cohort that evaluated AZD9291 treatment in combination with MEDI4736 as 1st line treatment has been terminated due to an increased incidence of ILD-like events (interstitial lung disease/pneumonitis), and is no longer being evaluated in this study.
  Other Names: Osimertinib & Durvalumab
  Arms: MEDI4736
Drug: Part C - AZD6094 monotherapy (Japan only) — Part C - AZD6094 monotherapy to assess the safety, tolerability and pharmacokinetics of the monotherapy of AZD6094 in Japanese patients with advanced NSCLC.
  Other Names: Savolitinib/Volitinib
  Arms: AZD6094 (monotherapy)
Drug: Part C - AZD9291 in combination with AZD6094 (Japan only) — Part C combination cohort - AZD9291 80mg OD administered in combination with AZD6094 400mg OD (AZD6094 dose in which DLTs have not been identified in the Japanese monotherapy cohort) in order to confirm the safety, tolerability, pharmacokinetics and preliminary anti-tumor activities of this combination in Japanese subjects. The 400mg OD dosing schedule will be initiated in the first cohort. The dose may be subsequently reduced in further cohorts in response to emerging safety, or PK findings or other reasons identified in the savolitinib programme.
  Other Names: Osimertinib & Savolitinib/Volitinib
  Arms: AZD6094
Drug: Part D - AZD9291 in combination with AZD6094 — Part D - AZD9291 80mg OD administered in combination with AZD6094 300mg OD to further evaluate the safety, tolerability, pharmacokinetics and antitumor activity in terms of ORR and PFS in patients with locally advanced or metastatic cMET positive EGFRm+ and T790M-negative NSCLC, following progression on EGFR-TKI treatment. The choice of AZD6094 dose of 300 mg is based on results from preclinical and clinical studies. Clinical testing of the 300 mg OD dose will enable better assessment of impact of lower AZD6094 exposure on overall tolerability and hepatotoxicity risk as well as exploration of the efficacy and overall safety profiles with a dose meaningfully lower than the current dose of 600 mg OD.
  Other Names: Osimertinib & Savolitinib/Volitinib
  Arms: AZD6094

SUMMARY:
The purpose of this study is to determine the safety, tolerability and preliminary anti-tumour activity of AZD9291 when given together with AZD6094 or selumetinib in patients with EGFR mutation positive advanced lung cancer

DETAILED DESCRIPTION:
This is a Phase Ib, open-label, multicentre study of AZD9291 administered orally in combination with novel therapeutics (AZD6094 or selumetinib (AZD6244, ARRY142886)) to patients with EGFRm+ advanced NSCLC. The study has been designed to allow an investigation of the optimal combination dose and schedule whilst ensuring the safety of patients with intensive safety monitoring. There are three main parts to this study; Part A, Combination dose finding and Parts B and D, Dose expansion. Part C, AZD6094 dose finding sub-study in advanced solid tumour patients is ongoing in Japan.

AZD9291 (osimertinib) is a potent irreversible inhibitor of both the single epidermal growth factor receptor sensitising mutation positive (EGFRm+) (tyrosine kinase inhibitor [TKI] sensitivity-conferring mutation) and dual EGFRm+/T790M+ (TKI resistance-conferring mutation) receptor forms of EGFR. AZD9291 therefore has the potential to provide clinical benefit to patients with advanced non-small cell lung cancer (NSCLC) harbouring both the single sensitivity mutations and the resistance mutation following prior therapy with an EGFR TKI. AZD9291 (osimertinib) was awarded FDA accelerated approval in November 2015, followed by conditional approval in the EU, full approval in Japan and additional markets in 2016, for the treatment of patients with EGFR T790M+ NSCLC who have progressed on or after EGFR TKI therapy.

Enrolment into the patient cohort that evaluated AZD9291 treatment in combination with MEDI4736 as 1st line treatment has been terminated due to an increased incidence of ILD-like events (interstitial lung disease/pneumonitis), and is no longer being evaluated in this study.

.

ELIGIBILITY:
Inclusion Criteria Signed informed consent Male or female aged at least 18 years and older. Patients from Japan aged at least 20 years.

Histological or cytological confirmation of EGFRm+ NSCLC. Confirmation that the tumour harbours an EGFR mutation known to be associated with EGFR TKI sensitivity (including exon 19 deletion and L858R). Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI eg, gefitinib or erlotinib. These patients must have radiological progression (as per site assessment) on the last treatment administered prior to enrolling in the study.

At least one lesion, not previously irradiated, not biopsied during the screening period, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with computerised tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements. Adequate haematological, liver and renal function as well as coagulation parameters.

ECOG/WHO performance status of 0 or 1 or KPS >80. Ability to swallow and retain oral medications. Prior to study entry, local confirmation of tumour cMET status is acceptable, a central result will be confirmed retrospectively. Local confirmation of tumour T790M status is acceptable if performed with an approved test and agreed by AstraZeneca.

Agree to use adequate contraceptive measures.

Exclusion Criteria Treatment with an EGFR TKI within approximately 5x half-life (eg, within 8 days for erlotinib, gefitinib or afatanib, or within 10 days for dacomitinib) of the first dose of study treatment. Any cytotoxic chemotherapy, investigational agents or other anticancer drugs for the treatment of advanced NSCLC from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment Patients currently receiving medications or herbal supplements known to be potent inducers of CYP3A4 (at least 3 weeks prior). For AZD6094 patients currently receiving prior to receiving the first dose, medications known to be strong inhibitors of CYP1A2.

Prior AZD9291 dosing in the present study. Prior treatment with a 3rd generation (T790M-directed) therapy (eg, AZD9291, rociletinib or HM61713) outside of this study is permitted if allocated to the 3rd generation EGFR TKI cohort. Prior or current treatment with AZD6094 or another cMET inhibitor (eg, foretinib, crizotinib, cabozantinib, onartuzumab) if allocated to AZD9291 plus AZD6094 combination. Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within ≥4 weeks of the first dose of study treatment Major surgical procedure, or significant traumatic injury within 4 weeks of the first dose of study treatment, or have an anticipated need for major surgery during the study.

Currently receiving treatment with warfarin sodium. LMWH is allowed. Active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy Any of the following cardiac diseases currently or within the last 6 months: Unstable angina pectoris, Congestive heart failure (NYHA ≥ Grade 2), Acute myocardial infarction, Stroke or transient ischemic attack.

Known hypersensitivity to the active or inactive excipients of AZD6094. Uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy) Mean resting correct QT interval (QTcF) >470 msec for women and >450 msec for men or factors that may increase the risk of QTcF prolongation such as chronic hypokalaemia not correctable with supplements, congenital or familial long QT syndrome, or family history of unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsade de Pointes.

Any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiograms (ECGs), e.g. complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec. Serious underlying medical condition at the time of treatment that would impair the ability of the patient to receive protocol treatment.

Active hepatitis B (positive HBsAg result) or hepatitis C (HCV). Patients with a past or resolved HBV infection are eligible if negative for HBsAg and positive for anti-HBc or positive for HBsAg, but for > 6 months have had normal transaminases and HBV DNA levels between 0-2000 IU/ml (inactive carrier state) and willing to start and maintain antiviral treatment for at least the duration of the study. HBV DNA levels > 2000 IU/ml but on prophylactic antiviral treatment for the past 3 months and will maintain the antiviral treatment during the study. Patients with positive HCV antibody are eligible only if the polymerase chain reaction is negative for HCV RNA.

Known serious active infection including, but not limited to, tuberculosis, or human immunodeficiency virus (positive HIV 1/2 antibodies).

Presence of other active cancers, or history of treatment for invasive cancer, within the last 5 years. Patients with Stage I cancer who have received definitive local treatment at least 3 years previously, and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.

Women who are either pregnant or breast feeding. Previous allogeneic bone marrow transplant Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events and/or Dose Limiting Toxicities as a Measure of Safety and Tolerability of AZD9291 when given in combination with AZD6094 or selumetinib | Adverse events will be collected from baseline until 28 days after the last dose in the AZD6094 or selumetinib arms.
  Part A: To investigate the safety and tolerability of AZD9291 when given in combination with AZD6094 or selumetinib who have progressed following prior therapy with an EGFR TKI agent, and define the combination dose(s) for further clinical evaluation.
Number of participants with Adverse Events as a measure of Safety and Tolerability of AZD9291 when given in combination with AZD6094 or selumetinib | Adverse events: baseline until 28 days after the last dose in the AZD6094 or selumetinib arms.
  Part B: To investigate the safety and tolerability of AZD9291 when given in combination with AZD6094 or selumetinib in patients with locally advanced or metastatic NSCLC, who have progressed on prior therapy with an EGFR TKI agent.
  Part C monotherapy cohort (Japan only): To investigate and confirm the safety and tolerability of AZD6094 when given orally to Japanese patients with advanced solid malignancies.
  Part C combination cohort (Japan only): To investigate the safety and tolerability of AZD9291 when given orally to Japanese patients with EGFRm+ NSCLC in combination with AZD6094 who have progressed following prior therapy with an EGFR TKI agent, and define the combination dose(s) for further clinical evaluation.
  Part D: To investigate the safety and tolerability of AZD9291 when given in combination with AZD6094 (300 mg OD) in patients with locally advanced or metastatic EGFRm+ NSCLC.

SECONDARY OUTCOMES:
Cmax after single dosing | Blood samples will be collected from each subject at pre-specified times on cycle 1 day 1 up to 24 hours
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
Tmax after single dosing | Blood samples will be collected from each subject at pre-specified on cycle 1 day 1 up to 24 hours
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
AUC after single dosing | Blood samples will be collected from each subject at pre-specified times on cycle 1 day 1 up to 24 hours
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
AUC0-t after single dosing | Blood samples will be collected from each subject at pre-specified on cycle 1 day 1 up to 24 hours
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
AUC0-24 after single dosing | Blood samples will be collected from each subject at pre-specified times on cycle 1 day 1 up to 24 hours
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
Terminal half life after single dosing | Blood samples will be collected from each subject at pre-specified times on cycle 1 day 1 up to 24 hours
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
CL/f after single dosing | Blood samples will be collected from each subject at pre-specified times on cycle 1 day 1 up to 24 hours
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
Volume of distribution after single dosing | Blood samples will be collected from each subject at pre-specified times on cycle 1 day 1 up to 24 hours
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
Cssmax after multiple dosing | Blood samples will be collected from each subject at pre-specified times on cycle 2 day 1 up to 24 hours
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
Tssmax after multiple dosing | Blood samples will be collected from each subject at pre-specified times on cycle 2 day 1 up to 24 hours
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
Cssmin after multiple dosing | Blood samples will be collected from each subject at pre-specified times for the duration of treatment.
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
AUCss after multiple dosing | Blood samples will be collected from each subject at pre-specified times on cycle 2 day 1 up to 24 hours
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
CLss/f after multiple dosing | Blood samples will be collected from each subject at pre-specified times on cycle 2 day 1 up to 24 hours
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
Rac after multiple dosing | Blood samples will be collected from each subject at pre-specified times on cycle 1 day 1 and cycle 2 day 1
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
Time dependency of PK after multiple dosing | Blood samples will be collected from each subject at pre-specified times on cycle 1 day 1 and cycle 2 day 1
  To characterise the pharmacokinetics of AZD9291, AZD6094 or selumetinib and metabolites after single dosing and at steady state after multiple dosing when AZD9291 is given orally in combination with AZD6094 or selumetinib (or, in case of Part C monotherapy for Japanese subjects, when AZD6094 is given alone) to patients with EGFRm+ NSCLC through plasma concentrations.
Objective response rate | At baseline and every 6 weeks until disease progression or withdrawal from study.
  To obtain a preliminary assessment of the anti-tumour activity of the combination of AZD9291 and AZD6094 or selumetinib by evaluation of tumour response (objective response rate, duration of response, change in tumour size) and progression free survival using RECIST version 1.1.
Disease control rate | At baseline and every 6 weeks until disease progression or withdrawal from study.
  To obtain a preliminary assessment of the anti-tumour activity of the combination of AZD9291 and AZD6094 or selumetinib by evaluation of tumour response (objective response rate, duration of response, change in tumour size) and progression free survival using RECIST version 1.1
Duration of response | At baseline and every 6 weeks until disease progression or withdrawal from study.
  To obtain a preliminary assessment of the anti-tumour activity of the combination of AZD9291 and AZD6094 or selumetinib by evaluation of tumour response (objective response rate, duration of response, change in tumour size) and progression free survival using RECIST version 1.1
Percentage change in tumour size | At baseline and every 6 weeks until disease progression or withdrawal from study.
  To obtain a preliminary assessment of the anti-tumour activity of the combination of AZD9291 and AZD6094 or selumetinib by evaluation of tumour response (objective response rate, duration of response, change in tumour size) and progression free survival using RECIST version 1.1
Progression free survival | At baseline and every 6 weeks until disease progression or withdrawal from study.
  To obtain a preliminary assessment of the anti-tumour activity of the combination of AZD9291 and AZD6094 or selumetinib by evaluation of tumour response (objective response rate, duration of response, change in tumour size) and progression free survival using RECIST version 1.1 Expansion phase only
Overall survival | Confirmed during the FUP period and at least every 12 weeks until the data cut-off for the primary analysis and determination that no further OS collection is needed, approximately 5 years, death, or full withdrawal of consent, whichever comes first.
  To obtain a preliminary assessment of overall survival in the AZD9291+AZD6094 combination arms of the study for Parts B and D.

CONTACTS AND LOCATIONS:
Overall Officials: Pasi A Jänne, MD, PhD, Principal Investigator — Dana-Faber Cancer Institute
Locations (31):
- United States (5):
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
- Canada (2):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
- Japan (5):
  - Research Site, Chūōku
  - Research Site, Habikino-shi
  - Research Site, Hirakata-shi
  - Research Site, Kashiwa
  - Research Site, Nagoya
- Poland (5):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
- Russia (5):
  - Research Site, Chelyabinsk
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Saint Petersburg
- South Korea (4):
  - Research Site, Cheongju-si
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taipei
- Ukraine (2):
  - Research Site, Kyiv
  - Research Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Ahn MJ, Cho BC, Ou X, Walding A, Dymond AW, Ren S, Cantarini M, Janne PA. Osimertinib Plus Durvalumab in Patients With EGFR-Mutated, Advanced NSCLC: A Phase 1b, Open-Label, Multicenter Trial. J Thorac Oncol. 2022 May;17(5):718-723. doi: 10.1016/j.jtho.2022.01.012. Epub 2022 Feb 15. PMID 35181499
- [Derived] Yoh K, Hirashima T, Saka H, Kurata T, Ohe Y, Hida T, Mellemgaard A, Verheijen RB, Ou X, Ahmed GF, Hayama M, Sugibayashi K, Oxnard GR. Savolitinib +/- Osimertinib in Japanese Patients with Advanced Solid Malignancies or EGFRm NSCLC: Ph1b TATTON Part C. Target Oncol. 2021 May;16(3):339-355. doi: 10.1007/s11523-021-00806-5. Epub 2021 May 3. PMID 33939068
- [Derived] Oxnard GR, Yang JC, Yu H, Kim SW, Saka H, Horn L, Goto K, Ohe Y, Mann H, Thress KS, Frigault MM, Vishwanathan K, Ghiorghiu D, Ramalingam SS, Ahn MJ. TATTON: a multi-arm, phase Ib trial of osimertinib combined with selumetinib, savolitinib, or durvalumab in EGFR-mutant lung cancer. Ann Oncol. 2020 Apr;31(4):507-516. doi: 10.1016/j.annonc.2020.01.013. Epub 2020 Jan 24. PMID 32139298
- [Derived] Sequist LV, Han JY, Ahn MJ, Cho BC, Yu H, Kim SW, Yang JC, Lee JS, Su WC, Kowalski D, Orlov S, Cantarini M, Verheijen RB, Mellemgaard A, Ottesen L, Frewer P, Ou X, Oxnard G. Osimertinib plus savolitinib in patients with EGFR mutation-positive, MET-amplified, non-small-cell lung cancer after progression on EGFR tyrosine kinase inhibitors: interim results from a multicentre, open-label, phase 1b study. Lancet Oncol. 2020 Mar;21(3):373-386. doi: 10.1016/S1470-2045(19)30785-5. Epub 2020 Feb 3. PMID 32027846